CLINICAL TRIAL: NCT05617261
Title: Evaluating Patient Tolerability and Success for Penile and Scrotal Urologic Procedures Under Conscious Sedation: A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, PremalPatel, Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education, University of Manitoba
Other Study IDs: HS25658 (B2022:092)
Record Dates: First submitted 2022-11-03; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Hydrocele; Spermatocele; Varicocele; Epididymal Cyst; Testicular Biopsy; Circumcision; Frenulectomy; Penile Plication; Orchiectomy; Vasectomy Reversal; Testicular Diseases; Penile Diseases
Keywords: Conscious sedation; Local anesthesia; Penile; Scrotal; Patient reported outcomes
MeSH Terms: conditions — Testicular Hydrocele; Spermatocele; Varicocele; Testicular Diseases; Penile Diseases | interventions — Conscious Sedation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Conscious sedation — Conscious sedation is a combination of medications to help you relax (a sedative, for example nitrous gas) and to block out pain (commonly known as freezing, for example lidocaine).

SUMMARY:
The goal of this observational study is to evaluate patient reported outcomes and tolerability of scrotal and penile urologic procedures under the administration of minimal conscious sedation. This will be assessed at 4-6 weeks post-procedure where patients will be followed up with a questionnaire assessing how well patients tolerated the procedure and if patients would opt for conscious sedation again in a similar, future procedure. The investigators will secondarily be assessing the associated cost savings as compared to having these procedures performed under general anesthesia at a tertiary care hospital.

DETAILED DESCRIPTION:
Background:

The current standard of care for the vast majority of urological procedures is the administration of general anesthesia, spinal anesthesia, or anesthesia-delivered sedation - requiring the operating room. However, this poses significant challenges associated with operating room costs, resources, and patient wait times. Given lengthy surgical backlogs, priority is focused on more acute conditions such as malignancies that require immediate intervention. Procedures for non-acute conditions, such as penile and scrotal procedures, have wait times that can exceed six months. Since most treatment for penile and scrotal cases tends to be surgical intervention, delays in these procedures may significantly negatively impact patients' sexual health, relationships, mental health, and quality of life. The ability to perform these procedures outside of the operating room using local anesthesia with or without conscious sedation may significantly reduce patient wait times and the costs of surgical intervention. Furthermore, the use of conscious sedation would allow for faster post-operative recovery, shorter procedural times, and decreased risks/side effects associated with general anesthesia.

Fields such as plastic surgery have successfully transitioned certain procedures into a clinic- based setting and the field of urology had also shown a similar interest. The investigators research team has been at the forefront of this transition - previously demonstrating the efficacy of distal ureteroscopy under nursing administered conscious sedation and other common urologic procedures. However, these studies were limited as they did not examine invasive scrotal and penile procedures, which have an extraordinary impact on the sexual health of patients.

Significance:

This project will provide evidence on the efficacy and characteristics of successful penile and scrotal procedures conducted under the administration of local anesthesia with or without conscious sedation. The findings of this study will help transition additional urological procedures into a clinic-based setting safely: improving the sexual and mental health of patients while decreasing cost, wait times, procedure duration, recovery times, and anesthetic-related complications.

Methods:

The proposed study is a prospective study. Eligible patients at the Manitoba Men's Health Clinic (Winnipeg, MB, Canada) will be approached for potential enrollment. Procedures with or without conscious sedation are routinely performed at this clinic with volumes of 15-20 procedures performed weekly.

Patients will be approached individually for potential recruitment into the study. Prior to their urological procedure, patients will be seen by a member of the research team to determine if they are willing to participate in the study. These meetings will occur in the pre-operative waiting room at the Manitoba Men's Health Clinic where a member of the research team who is involved in the care of that patient, will review the medical chart to ensure the candidate meets the inclusion and exclusion criteria of the study. After discussing the study, potential participants will have the opportunity to decide whether they would like to be involved or not. Those who choose to be involved in the study will have to sign an informed consent form. Patients may withdraw consent and terminate participation at any time.

Each participant will be assigned a study number to track them over time. Electronic data forms will be used to collect preliminary information for all patients who consent to the study. Baseline variables for collection will include patient age, sex, BMI, co-morbidities, medications, smoking/drinking/illicit substance use, and family history of notable diseases. Clinical variables collected will include procedure side (where applicable), medication dose used for sedation, quantity and type of local anesthetic, procedural and recovery times, patient-reported and surgeon-reported visual analogue scale pre-, intra-, and post-operation.

The statistical tests will include univariable and multivariable analyses. All the variables defined above in the data collection section will be analyzed to determine if there is an association between any of these variables and the patient-reported outcomes after the urological procedure. Normally distributed continuous data will be reported as the mean ± the standard deviation. Non-normally distributed data will be presented using the median and the interquartile range. Multivariable adjusted logistic regression analysis will be used to assess predictors of whether a patient would opt for conscious sedation again as opposed to general/spinal anesthesia. SPSS Version 24.0 (SPSS Inc, IBM, Chicago, IL) will be used for data analysis.

Personal Health Information Act (PHIA) compliance of the investigators database will be ensured by preventing unauthorized access and implementing security measures such as password protecting the electronic database and never permanently storing the database on a mobile device or flash drive. Data will only be stored on the desktop computer enclosed in the Manitoba Men's Health Clinic. Database information will only be emailed using a password- protected, encrypted file. Information presented at meetings and conferences will be de- identified and anonymous. The Research Ethics Board has approved this study at the University of Manitoba.

ELIGIBILITY:
Inclusion Criteria:

1. patients over the age of 18
2. undergoing one of the previously mentioned procedures under local anesthesia with or without conscious sedation
3. having a minimum follow-up of 4-6 weeks.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing: hydrocelectomy, spermatocelectomy, varicocelectomy, epididymectomy, testicular biopsy, adult circumcision, frenulectomy, penile plication, orchiectomy, and vasectomy reversal at the Manitoba Men's Health Clinic (Winnipeg, MB, Canada) will be approached for potential enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-13 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported tolerability | Standardized questionnaire will be administered to patients 4-6 weeks after their individual procedure.
  Patient tolerability as assessed using a standardized questionnaire administered to patients. Key questions of interest are if patients would opt for conscious sedation for a repeat procedure or general anesthesia, recommend conscious sedation to a friend undergoing a similar procedure, and a scale question with self-reported tolerability ranging from 0-10 with a higher value corresponding to an excellent experience.

CONTACTS AND LOCATIONS:
Overall Officials: Premal Patel, MD, Principal Investigator — Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education
Locations (1):
- Men's Health Clinic Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Bal DS, Chung D, Urichuk M, Shah J, Fidel MG, Panchendrabose K, Sidhom K, Bard R, Nayak JG, Patel P. Utilizing Local Anesthesia Only for Penile and Scrotal Urologic Surgery: A Prospective Study on Patient Tolerability and Surgical Outcomes for a Sedation-free Option. Urology. 2024 Dec;194:7-13. doi: 10.1016/j.urology.2024.08.051. Epub 2024 Aug 28. PMID 39208947